CLINICAL TRIAL: NCT04630769
Title: Intraperitoneal FATE FT516 and Interleukin-2 (IL-2) With Intravenous Enoblituzumab in Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: FT516 and IL2 With Enoblituzumab for Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020LS001; P01CA111412 (NIH)
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer; Fallopian Tube Adenocarcinoma; Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Interleukin-2

STUDY DESIGN:
Intervention Model Description: This study is conducted in two consecutive stages with 5 cohorts. A minimum of 28 days must separate each cohort. Within a 3 patient cohort, a minimum of 14 days must separate the first and second patient. Stage 1 Step 1 uses a fast-track design (1 patient per cohort) with a minimum of 28 days between each patient until one of the following: a) 1st occurrence of a pre-defined adverse event at which point the study moves to Step 2. The cohort size increases from 1 to 3 patients with 2 additional patients added. Escalation in Step 2 continues until the 1st DLT at which point Stage 2 continual reassessment method (CRM) is activated. If Cohort 5 is completed with 10 patients enrolled at the MTD without a DLT, Stage 2 (CRM) is not used. b) The 1st occurrence of a DLT the study moves directly to Stage 2 (CRM) and Step 2 is not used. c) Cohort 5 is completed without a pre-defined AE or a DLT - neither Step 2 nor Stage 2 is used if a total of 10 patients are enrolled in Cohort 5.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Monotherapy: IP FT516 at 9 x 10^7 cells/dose on Day 1, 8, and 15 (Experimental)
  Interventions: Drug: IP FT516; Drug: IL-2
- Monotherapy: IP FT516 at 3 x 10^8 cells/dose on Day 1, 8, and 15 (Experimental)
  Interventions: Drug: IP FT516; Drug: IL-2
- Monotherapy: IP FT516 at 9 x 10^8 cells/dose on Day 1, 8, and 15 (Experimental)
  Interventions: Drug: IP FT516; Drug: IL-2
- Safe dose (MTD-1) from 1st 3 levels + IV enoblituzumab on Day -6 (Experimental)
  Interventions: Drug: IP FT516; Drug: Enoblituzumab; Drug: IL-2
- Highest dose (MTD) from 1st 3 levels + IV enoblituzumab on Day -6 (Experimental)
  Interventions: Drug: IP FT516; Drug: Enoblituzumab; Drug: IL-2

INTERVENTIONS:
Drug: IP FT516 — FT516 is an off-the-shelf cryopreserved NK cell product derived from an iPSC that was transduced with a high affinity, ADAM17 non-cleavable CD16 (Fc receptor) that maintains CD16 on the cell surface, which remains fully functional after NK cell activation
Drug: Enoblituzumab — Enoblituzumab is an Fc-optimized monoclonal antibody that targets B7-H3 which is highly expressed on ovarian cancer. Enoblituzumab at 15 mg/kg IV, one day before lymphodepleting chemotherapy
  Arms: Highest dose (MTD) from 1st 3 levels + IV enoblituzumab on Day -6; Safe dose (MTD-1) from 1st 3 levels + IV enoblituzumab on Day -6
Drug: IL-2 — IL-2 at 6 Million IU (3 Million IU/m2 if patient weight is <45 kg) is administered IP in 50 cc of room temperature D5W via peritoneal catheter directly after the FT-516 infusion is completed. Immediately following the IL-2, an additional 100 cc D5W flush is infused into the peritoneal cavity through the peritoneal catheter as rapidly as possible.
  Other Names: Interleukin-2

SUMMARY:
This is a single center Phase I clinical trial of FT516 administered intraperitoneally (IP) once a week for 3 consecutive weeks for the treatment of recurrent gynecologic cancers. As this is an early 1st in human study and the 1st intraperitoneal infusion of FT516, the safety of FT516 is confirmed prior to adding enoblituzumab as an intravenous infusion approximately 1 week prior to the 1st dose of FT516 and every 3 weeks beginning on Day 22 (1 week after the last dose of FT516). Each dose of FT516 is followed directly by an IP infusion of interleukin-2 (IL-2) to facilitate natural killer (NK) cell survival. A short course of outpatient lymphodepletion chemotherapy is given prior to the 1st dose of FT516.

DETAILED DESCRIPTION:
FT516 is an off the shelf product comprised of allogeneic natural killer (NK) cells, expressing high-affinity non-cleavable CD16 (FT516). Enoblituzumab is an Fc-optimized monoclonal antibody that targets B7-H3 which is highly expressed on ovarian cancer. Based on data showing that within the ovarian cancer tumor microenvironment surface expression of CD16a on NK cells is diminished, the researchers hypothesize that the FT516 cellular product containing a non-cleavable CD16 will bypass the low CD16 expression issue and maximize NK cell cytotoxicity. Enoblituzumab is an Fc optimized humanized IgG1 monoclonal antibody that binds to B7-H3 (CD276). B7-H3 is an inhibitory immune checkpoint molecule that is widely expressed by a number of different tumor types and may play a key role in regulating the immune response. It is therefore hypothesized that the combination of FT516 with enoblituzumab will maximize NK cell cytotoxicity in patients with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer meeting one of the following minimal prior treatment requirement (no limit to the maximum number of prior treatments):
* Platinum Resistant: may receive FT516 as 2nd line (as 1st salvage therapy) with platinum resistant is defined as disease that has responded to initial chemotherapy but demonstrates recurrence within a relatively short period of time (< 6 months) following the completion of treatment.
* Platinum Sensitive: may receive FT516 as 3rd line therapy (as 2nd salvage therapy) with platinum sensitive is defined as the recurrence of active disease in a patient who has achieved a documented response to initial platinum-based treatment and has been off therapy for an extended period of time (≥ 6 months).
* Measurable disease per modified Response Evaluation Criteria in Solid Tumors, v1.1 within the abdomen and pelvis assess within 42 days of the 1st FT516 infusion. Extra-peritoneal disease is permitted; however each lesion must be < 5 cm at the largest diameter.
* At least 18 years of age
* GOG Performance Status 0, 1, or 2
* Adequate organ function within 14 days of study registration (28 days for pulmonary and cardiac) defined as:
* Hematologic: platelets ≥ 75,000 x 10^9/L and hemoglobin ≥ 9 g/dL, unsupported by transfusions; absolute neutrophil count (ANC) ≥ 1000 x 10^9/L, unsupported by G-CSF or granulocytes
* Creatinine: Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m^2 per current institutional calculation formula
* Hepatic: AST and ALT ≤ 3 x upper limit of institutional normal
* Pulmonary Function: Oxygen saturation ≥ 90% on room air; PFT's required only if symptomatic or prior known impairment - must have pulmonary function >50% corrected DLCO and FEV1
* Cardiac Function: LVEF ≥ 40% by echocardiography, MUGA, or cardiac MRI; no clinically significant cardiovascular disease including any of the following: stroke or myocardial infarction within 6 months prior to first study treatment; unstable angina or congestive heart failure of New York Heart Association Grade 2 or higher
* Agrees to the placement of an intraperitoneal catheter before the 1st dose of study directed drug (chemotherapy or enoblituzumab - Cohort 4 and 5) and remains in place through Day 36 or longer if retreatment is planned
* Agrees to undergo a tumor biopsy if feasible at the time the catheter is placed and removed - Accessible tumor for biopsy is not required for eligibility.
* Washout period of at least 14 days after any standard of care tumor directed therapy prior to the first dose of investigational product (FT516 for Levels 1-3 or enoblituzumab for Levels 4-5)
* If history of brain metastases must be stable for at least 3 months after treatment - A brain CT scan or MRI is only be required in subjects with known brain metastases at the time of enrollment or in subjects with clinical signs or symptoms suggestive of brain metastases
* Must agree to and sign the consent for the companion Long-Term Follow-Up study (CPRC #2020LS072) to fulfill the FDA required 15 years of follow-up for a genetically modified cell product
* Voluntary written consent prior to the performance of any research related procedures

Exclusion Criteria:

* Pregnant or breastfeeding or planning on becoming pregnant in the next 6 months. Woman of childbearing potential who still have a uterus and ovaries, must agree to use at effective contraception and must have a negative pregnancy test within 14 days of study enrollment.
* Any known condition that requires systemic immunosuppressive therapy (> 5mg prednisone daily or equivalent) during the FT516 dosing period (3 days before the 1st dose through 14 days after the last dose) - topical and inhaled steroids are permitted.
* Active autoimmune disease requiring systemic immunosuppressive therapy
* History of severe asthma and currently on chronic systemic medications (mild asthma requiring inhaled steroids only is eligible)
* Uncontrolled bacterial, fungal or viral infections with progression of clinical symptoms despite therapy
* Receipt of any investigational agent within 28 days prior to the first dose of investigational product (FT516 for Levels 1-3 or enoblituzumab for Levels 4-5)
* Live vaccine <6 weeks prior to start of lympho-conditioning
* Known allergy to the following FT516 components: albumin (human) or DMSO
* Any history of prior enoblituzumab administration
* Known history of HIV positivity or active hepatitis C or B - chronic asymptomatic viral hepatitis is allowed
* Presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, MS, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15 | Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6 | Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6
Started | 1 | 1 | 1 | 0 | 0
Completed | 1 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in 'Safe dose (MTD-1) from 1st 3 levels + IV enoblituzumab on Day -6' or 'Highest dose (MTD) from 1st 3 levels + IV enoblituzumab on Day -6 ' Arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15 | Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6 | Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  |  | 0
  Between 18 and 65 years | 1 | 1 | 1 |  |  | 3
  >=65 years | 0 | 0 | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 |  |  | 3
  Male | 0 | 0 | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 |  |  | 0
  Not Hispanic or Latino | 1 | 1 | 1 |  |  | 3
  Unknown or Not Reported | 0 | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  |  | 0
  Asian | 0 | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 | 0 |  |  | 0
  White | 1 | 1 | 1 |  |  | 3
  More than one race | 0 | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicity (DLT) Events
Description: DLT is defined as any treatment emergent toxicity at least possibly related to the study treatment meeting one of the following criteria based on CTCAE v5 within 28 days (14 days for ascites) of the 1st FT516 infusion (for Cohort 4 and 5, DLT assessment starts with enoblituzumab and continues for 28 days after 1st FT516): Grade 3 organ toxicity (pulmonary, hepatic, renal, or neurologic) not pre-existing and lasting more than 72 hours , Any non-hematologic Grade 4 or 5 toxicity, Neutrophil count decreased ≥ Grade 4 that persists at Day 28 despite use of growth factor support ,Grade 3 abdominal pain lasting more than 4 consecutive days and not controlled by standard analgesics, Grade 3 or greater ascites within 14 days after FT516 administration in patients who had no ascites or Grade 1 ascites at enrollment and is not attributable to disease progression
Time Frame: 28 Days Post FT516 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15
Number analyzed (Participants) | 1 | 1 | 1
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing adverse events related to FT516
Time Frame: 28 days after first dose of FT516 or 28 days after last dose of Enoblituzumab (arm 4 and 5 only)
Population: No participants were enrolled in the "Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6" and "Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6" arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15
Number analyzed (Participants) | 1 | 1 | 1
Participants | 1 | 1 | 1

3. Secondary Outcome: Number of Participants Experiencing Progression Free Survival
Description: Number of participants experiencing progression free survival at 6 months from the first dose of FT516
Time Frame: 6 months from the first dose of FT516
Population: No data collected as no participants were on study at 6 months from first dose of FT516 in the "Monotherapy: IP FT516 at 9 x 10^7 cells/dose on Day 1, 8, and 15" and "Monotherapy: IP FT516 at 9 x 10^8 cells/dose on Day 1, 8, and 15" arms.
  No data collected as no participants were enrolled in the "Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6" and "Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6" arms.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6; Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6: IP FT516: FT516 is an off-the-shelf cryopreserved NK cell product derived from an iPSC that was transduced with a high affinity, ADAM17 non-cleavable CD16 (Fc receptor) that maintains CD16 on the cell surface, which remains fully functional after NK cell activation
  IL-2: IL-2 at 6 Million IU (3 Million IU/m2 if patient weight is <45 kg) is administered IP in 50 cc of room temperature D5W via peritoneal catheter directly after the FT-516 infusion is completed. Immediately following the IL-2, an additional 100 cc D5W flush is infused into the peritoneal cavity through the peritoneal catheter as rapidly as possible.
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15 | Experimental: Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6 | Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 0
Participants | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Experiencing Progression Free Survival
Description: Number of participants experiencing progression free survival at 1 year from the first dose of FT516
Time Frame: 1 year from the first dose of FT516
Population: No data collected as no participants were enrolled in the "Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6" and "Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6" arms.
  No data collected as no participants were on study at 1 year from first dose of FT516 for all remaining arms.
Measure: Number; unit: Participants
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15 | Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6 | Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 0
Participants | 0 | 0 | 0 |  |

5. Secondary Outcome: Number of Participants Experiencing Overall Survival
Description: Number of participants experiencing overall survival at 6 months from the first dose of FT516
Time Frame: 6 months from the first dose of FT516
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15
Number analyzed (Participants) | 1 | 1 | 1
Participants | 0 | 1 | 0

6. Secondary Outcome: Number of Participants Experiencing Overall Survival
Description: Number of participants experiencing overall survival at 1 year from the first dose of FT516
Time Frame: 1 year from the first dose of FT516
Population: as for outcome 4
Measure: Number; unit: Count of Participants
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15 | Safe Dose (MTD-1) From 1st 3 Levels + IV Enoblituzumab on Day -6 | Highest Dose (MTD) From 1st 3 Levels + IV Enoblituzumab on Day -6
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 0
Count of Participants | 0 | 0 | 0 |  |

ADVERSE EVENTS:
Time Frame: Adverse events were assessed through day 28 after the 1st dose of FT516. After day 28, All-Cause Mortality was assessed up to approximately 9 months from the first dose of FT516.
Arm/Group | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 (N=1) | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 (N=1) | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15 (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monotherapy: IP FT516 at 9 x 10^7 Cells/Dose on Day 1, 8, and 15 (N=1) | Monotherapy: IP FT516 at 3 x 10^8 Cells/Dose on Day 1, 8, and 15 (N=1) | Monotherapy: IP FT516 at 9 x 10^8 Cells/Dose on Day 1, 8, and 15 (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (6) | 1 (3) | 1 (4)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (4) | 1 (11)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (4) | 1 (4)
Vomiting (Gastrointestinal disorders) | 1 (5) | 1 (2) | 1 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1) | 1 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (4)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (4) | 1 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (8) | 1 (9) | 1 (6)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (3) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (5) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT04630769/Prot_SAP_000.pdf